## Sustainable Football: Physical Profile, Training Load, Risk Factors and Injuries in Swedish Elite Football

Date: 2024-07-28

## Data analysis and statistics

Statistics will be computed using IBM SPSS Statistics (New York, USA). To compare means between the groups (academy vs professional players, injured vs non-injured players, men vs women), independent student T-tests will be used. The binary logistic regression will be used to verify whether different levels of physical performance have impact on the risk of injury. The one-way ANCOVA, with Bonferroni correction for adjustment of multiple comparisons, will be used to analyze difference in adjusted means of test results between groups. Due to the explorative nature of the study and cohort design no sample size calculation will be performed.